CLINICAL TRIAL: NCT06420778
Title: A Randomized Controlled Study on the Treatment of Postherpetic Neuralgia in the Head and Face With Superficial Needling Combined With Electroacupuncture
Brief Title: The Treatment of Postherpetic Neuralgia in the Head and Face With Superficial Needling Combined With Electroacupuncture
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang Chinese Medical University (Other Government)
Responsible Party: Principal Investigator, Xiaoyu Li, Director, Zhejiang Chinese Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023ZR030
Record Dates: First submitted 2024-05-14; First posted 2024-05-20 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2024-06

CONDITIONS: Postherpetic Neuralgia; Electroacupuncture; Infrared Thermography
MeSH Terms: conditions — Neuralgia, Postherpetic | interventions — Electroacupuncture; Pregabalin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- therapy group (Experimental): Subjects in this group will be treated with Cluster needle shallow stabbing combined with electroacupuncture.The treatment time was 60 minutes each time, once every other day, and the treatment was carried out 3 times a week for 4 consecutive weeks, for a total of 12 treatments.
  Interventions: Other: electroacupuncture
- Control group (Experimental): Subjects in this group will be treated with oral pregabalin capsules only, 150 mg twice daily for 4 weeks.Pregabalin was administered with Lerica (specification: 75 mg*8 capsules,manufactured by Pfizer Pharmaceuticals Ltd).
  Interventions: Drug: Pregabalin

INTERVENTIONS:
Other: electroacupuncture — The patient takes the supine position, the whole body relaxes, the facial skin is routinely sterilized. Local acupuncture points along the head and face herpes zoster lesion branches with 0.18 × 25 mm millimetre needle series of shallow stabbing method row stabbing method.Han's Acupoint Neurostimulator (model HANS-200) was selected, local acupoints were chosen as Xiaguan+Quanliao or Xiaguan+Jiache, and distal acupoints were chosen as Hegu+Waiguan connected with electroacupuncture, sparse and dense wave 2/100 Hz was selected, and the treatment time was 60 minutes, and the intensity of the current was all to the extent that the patient could tolerate it. The needles were left in place for 60 minutes each time, once every other day, and the treatment was performed 3 times a week for 4 weeks, for a total of 12 treatments.
  Arms: therapy group
Drug: Pregabalin — Subjects in this group will be treated with oral pregabalin capsules only, 150 mg twice daily for 4 weeks.Pregabalin was administered with Lerica (specification: 75 mg*8 capsules,manufactured by Pfizer Pharmaceuticals Ltd).
  Arms: Control group

SUMMARY:
Based on the inclusion and exclusion criteria, patients with head and face PHN who met the requirements were selected as trial subjects, and the efficacy was clarified in a randomized controlled design trial. The visual analog score VAS was used as the primary evaluation index, and the depression self-assessment scale score , Hamilton depression scale, Pittsburgh sleep quality index scale, and quality of life evaluation scale (SF-36) were used as the secondary evaluation indexes, and oral pregabalin was used as the control group, and the subjects in the pregabalin and the plexus superficial stabbing combined with electroacupuncture groups were observed respectively at the time of Before treatment, immediately after the first treatment, after 2 days of treatment, after 2 weeks of treatment, after 4 weeks of treatment, after 1 month of follow-up after the end of treatment and after 2 months of follow-up after the end of treatment.

DETAILED DESCRIPTION:
On the one hand, it was clarified whether plexus needle shallow stabbing combined with electroacupuncture for the treatment of PHN in the head and face has clear and stable advantages in pain reduction, improvement of mood, sleep quality and quality of life, and formed the clinical standardization of plexus needle shallow stabbing combined with electroacupuncture for the treatment of postherpetic neuralgia in the head and face, which in turn lays the foundation for the further popularization of acupuncture for the treatment of postherpetic neuralgia in the head and face, and also provides a new, scientific and effective way of thinking about clinical analgesic therapies for postherpetic neuralgia.

On the other hand, this study will clarify the correlation between facial thermal radiation characteristics and clinical symptoms in patients with head and face PHN, and apply infrared thermography as an objective evaluation of the efficacy index of plexus needling and shallow stabbing combined with electroacupuncture in the treatment of head and face PHN, which will provide a new method for objectively verifying the clinical efficacy of PHN.

ELIGIBILITY:
Inclusion Criteria:

Meet the diagnostic criteria in the 2016 Chinese Expert Consensus on the Diagnosis and Treatment of Postherpetic Neuralgia; Age 50-80 years (including telangiectasia), gender is not limited; Have a history of herpes zoster on the head and face, and the lesions on the head and face have been healed and subsided, and the symptoms of neuralgia lasted ≥1 month after lesions were healed, with baseline scores of ≥4 on the Facial Pain Profile, and abnormal sensation of the skin around the lesions, pain sensitivity; Be conscious and have a clear sense of pain and discriminative ability; Sign the informed consent to participate in this study voluntarily. Only those who satisfy the above 5 items at the same time can be included in this study.

Exclusion Criteria:

those who did not meet the above diagnostic criteria; herpes zoster occurring in the perineum, or special types such as visceral herpes zoster, meningeal herpes zoster, and generalized herpes zoster; those who were taking oral pregabalin at a dose of less than 0.2 g or more than 0.6 g per day before inclusion to relieve analgesia; those who had a serious adverse reaction to pregabalin, were allergic to acupuncture, or belonged to patients who were within the range of contraindications to electro-acupuncture; Combined with severe cardiac, hepatic, renal damage, epilepsy, head injury, or cognitive dysfunction, aphasia, psychiatric disorders, and other major diseases, who are unable to cooperate with the treatment; Combined with poorly controlled hypertension and diabetes mellitus patients; Pregnant or breastfeeding patients;8.Patients who are currently participating in other studies, and who have been enrolled in other clinical trials within the last 3 months. Anyone who meets any of these criteria will be excluded.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2024-07-12 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale/Score | VAS will be performed at the baseline (pre-treatment), the 2 week after intervention,the 1 month after intervention,the 1 month follow-up and the 2 month follow-up to evaluate the severity of the disease and the treatment effect.
  This scale is performed by two trained raters to perform a Self-rating depression scale（SDS）, usually in the form of conversation and observation. After the examination, the two raters will score independently.Baseline values were taken from the pre-treatment assessment, mean values from weeks 1 and 2 of the treatment period were taken at mid-treatment (2 weeks), and mean values from weeks 3 and 4 of the treatment period were taken at the end of treatment (4 weeks). Daily mean values were taken for one month at one month follow-up and for two months at two months follow-up.

SECONDARY OUTCOMES:
Self-rating depression scale | SDS will be performed at the baseline (pre-treatment), the 2 week after intervention,the 1 month after intervention,the 1 month follow-up and the 2 month follow-up to evaluate the severity of the disease and the treatment effect.
  This scale is performed by two trained raters to perform a Self-rating depression scale（SDS）, usually in the form of conversation and observation. After the examination, the two raters will score independently.
Hamilton depression scale | HAMD will be performed at the baseline (pre-treatment), the 2 week after intervention,the 1 month after intervention,the 1 month follow-up and the 2 month follow-up to evaluate the severity of the disease and the treatment effect.
  This scale is performed by two trained raters to perform a Hamilton depression scale (HAMD), usually in the form of conversation and observation. After the examination, the two raters will score independently.
Pittsburgh Sleep Quality Index Scale | PSQI will be performed at the baseline (pre-treatment), the 2 week after intervention,the 1 month after intervention,the 1 month follow-up and the 2 month follow-up to evaluate the severity of the disease and the treatment effect.
  This scale is performed by two trained raters to perform a Pittsburgh Sleep Quality Index Scale（PSQI）, usually in the form of conversation and observation. After the examination, the two raters will score independently.
Quality of Life Rating Scale | SF-36 will be performed at the baseline (pre-treatment), the 2 week after intervention,the 1 month after intervention,the 1 month follow-up and the 2 month follow-up to evaluate the severity of the disease and the treatment effect.
  This scale is performed by two trained raters to perform aQuality of Life Rating Scale（SF-36）, usually in the form of conversation and observation. After the examination, the two raters will score independently.

CONTACTS AND LOCATIONS:
Locations (1):
- Xiaoyu Li, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Qiu P, Sun H, Xia Y, Qu S, Fang J, Li X. The efficacy of electroacupuncture for postherpetic neuralgia arising from herpes zoster affecting the cephalo-facial area: study protocol for a double center randomized controlled trial. Front Med (Lausanne). 2025 Aug 28;12:1616035. doi: 10.3389/fmed.2025.1616035. eCollection 2025. PMID 40950954